CLINICAL TRIAL: NCT00082589
Title: A Randomized, Double-Blind, Multi-Center,Study Evaluating the Effects of Eplerenone Versus Placebo on Ventricular Remodeling in Patient's With Left Ventricular Systolic Dysfunction (EF Less Than or Equal to 35%) and Mild to Moderate Heart Failure
Brief Title: The Purpose of This Study is to Determine if Eplerenone is Effective in Treatment of Mild to Moderate Heart Failure
Acronym: REMODEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A6141078
Record Dates: First submitted 2004-05-12; First posted 2004-05-14 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
The purpose of this study is to determine if eplerenone is effective in the treatment of mild to moderate heart failure

ELIGIBILITY:
Inclusion Criteria:

* Current symptoms consistent with mild to moderate heart failure (NYHA functional class II and III)
* LVEF (left ventricular ejection fraction) of <35% by equilibrium-gated RVG at screening
* Therapy with an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) and beta-blocker (BB) (unless documented intolerance) for at least 3 months duration and at dose that has not been adjusted within the previous 4 weeks

Exclusion Criteria:

* Current decompensated heart failure or heart failure hospitalization or severe heart failure (NYHA functional class IV) within 6 months of screening
* Use of eplerenone or spironolactone within 30 days of randomization or for more than 7 days within the previous 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-04; Study Completion 2006-03

PRIMARY OUTCOMES:
Difference between eplerenone and placebo in change from baseline in LV end diastolic volume index (EDVi) determined by equilibrium-gated radionuclide ventriculography (RVG)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (45):
  - Pfizer Investigational Site, Castro Valley, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Covington, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Bloomington, Illinois
  - Pfizer Investigational Site, Normal, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lexington, Nebraska
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, McCook, Nebraska
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, West Islip, New York
  - Pfizer Investigational Site, Mount Airy, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Lorain, Ohio
  - Pfizer Investigational Site, Sandusky, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Sayre, Pennsylvania
  - Pfizer Investigational Site, Pawtucket, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Galax, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Udelson JE, Feldman AM, Greenberg B, Pitt B, Mukherjee R, Solomon HA, Konstam MA. Randomized, double-blind, multicenter, placebo-controlled study evaluating the effect of aldosterone antagonism with eplerenone on ventricular remodeling in patients with mild-to-moderate heart failure and left ventricular systolic dysfunction. Circ Heart Fail. 2010 May;3(3):347-53. doi: 10.1161/CIRCHEARTFAILURE.109.906909. Epub 2010 Mar 18. PMID 20299607
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141078&StudyName=The+Purpose+of+this+Study+is+to+Determine+if+Eplerenone+is+Effective+in+Treatment+of+Mild+to+Moderate+Heart+Failure